CLINICAL TRIAL: NCT02685384
Title: Post ACA Reform: Evaluation of Community Health Center Care of Diabetes
Acronym: PREVENTD
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: OCHIN, Inc. (Other); Health Choice Network (Other); Fenway Community Health (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jennifer E DeVoe, MD DPhil, Associate Professor, Oregon Health and Science University
Other Study IDs: U18DP006116 (NIH)
Record Dates: First submitted 2016-02-04; First posted 2016-02-18 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus (DM)
Keywords: healthcare access; healthcare utilization; health expenditures; preventive services; biomarkers
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Medicaid Expansion States: Patients receiving care in community health centers in states that expanded Medicaid (intervention group)
  Interventions: Other: Medicaid Expansion
- Non Medicaid Expansion States: Patients receiving care in community health centers in states that did not expand Medicaid (control group)
  Interventions: Other: Medicaid Expansion

INTERVENTIONS:
Other: Medicaid Expansion — There will be no direct intervention, but rather an observation of change based on whether a state expanded Medicaid or not

SUMMARY:
This innovative and timely study will measure the impact of Affordable Care Act (ACA) Medicaid expansions on diabetes mellitus (DM) prevention, treatment, expenditures and health outcomes. To assess this natural policy experiment, the investigators will use electronic health record data from the ADVANCE clinical data research network (CDRN) of the National Patient-Centered Clinical Research Network (PCORnet).

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is one of the most prevalent chronic diseases, affecting over 29 million people in the United States (US). The number of people with DM is expected to increase by 200% between 2005 and 2050, from 16 to 48 million. Health insurance and continued access to healthcare services are essential for optimal DM care and management; thus, it is hypothesized that Affordable Care Act (ACA) Medicaid expansions could substantially improve access to health insurance and essential healthcare services for patients with DM risk (aged ≥45 + overweight) and patients diagnosed with DM. Studies of single state Medicaid expansions showed increased utilization of healthcare services, access to providers, receipt of preventive care services, and improved health outcomes post-expansion; however, past studies did not have concurrent control states. In 2012, the US Supreme Court ruled that states were not legally required to implement ACA Medicaid expansion, creating a 'natural policy experiment' - a unique national opportunity to test the effect of ACA Medicaid expansion on healthcare access and services for patients at risk for DM or diagnosed with DM ('with DM risk or DM'). By January 1, 2015, 28 states and the District of Columbia had implemented the expansion; Medicaid enrollment increased by an estimated 12.9% in expansion states, compared to 2.6% in non-expansion states. The investigators propose to use this unprecedented natural policy experiment to study the effect of state-level Medicaid expansions on DM prevention, treatment, expenditures, and health outcomes. As many persons affected by both DM and the ACA Medicaid expansions receive primary care in safety net community health centers (CHCs), the proposed analyses will use electronic health record (EHR) data from the national ADVANCE clinical data research network (CDRN) of CHCs (ADVANCE is one of 11 CDRNs in the national PCORnet data network). The ADVANCE CDRN has patient-level data from 470 CHCs in 12 Medicaid expansion states (n=1,242,823 patients) and 248 CHCs in 9 non-expansion states (n=830,399 patients). This nationally unique data resource will let the investigators measure pre-post DM-related utilization and receipt of preventive services in expansion versus non-expansion states, illuminating the impact of ACA Medicaid expansions on DM prevention and treatment Our proposed study, Post ACA Reform: EValuation of community hEalth ceNTer care of Diabetes (PREVENT-D) has the following specific aims:

Aim 1. Compare pre-post insurance status, overall visits, and chronic disease management visits among patients with DM risk or DM, in expansion versus non-expansion states.

Aim 2. Compare pre-post receipt of primary and secondary DM preventive services (e.g., screening for obesity, lipid levels, glycosylated hemoglobin) among patients with DM risk or DM, in expansion versus non-expansion states.

Aim 3. Compare pre-post changes in DM-related biomarkers (e.g., body mass index, blood pressure, lipid levels) in patients with DM risk or DM among newly insured (gained Medicaid in post-period), already insured (had coverage in pre- and post-period), and continuously uninsured (no coverage in pre- and post-period) patients in states that expanded Medicaid.

Aim 4: Measure pre-post changes in Oregon Medicaid expenditures among newly insured compared to already insured patients with DM risk or DM.

ELIGIBILITY:
Inclusion Criteria:

* Patients in intervention and control states aged 20-64

Exclusion Criteria:

* Patients at intervention and control clinics outside of the age range 20-64 Pregnant women to eliminate the possibility of having gestational diabetes mellitus diagnoses

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study eligible patients within electronic health record data from the ADVANCE clinical data research network (CDRN) of PCORnet
Sampling Method: Non-Probability Sample
Enrollment: 1938375 (Actual)
Dates: Start 2012-01; Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Change of health insurance status | 24 months prior to Medicaid expansion vs 24 months post
  Health insurance status derived from EHR data and is primarily based on information collected at each visit

SECONDARY OUTCOMES:
Change in number of internal services utilization | 24 months prior to Medicaid expansion vs 24 months post
  Number of internal services utilized including number and ratio of "traditional" face to face visits vs. "nontraditional" encounters and communication via phone, personal health record, and email
Change in type of internal services utilization | 24 months prior to Medicaid expansion vs 24 months post
  Type of internal services utilized including number and ratio of "traditional" face to face visits vs. "nontraditional" encounters and communication via phone, personal health record, and email
Change in number of preventive services received | 24 months prior to Medicaid expansion vs 24 months post
  Number of all billed encounters overall and yearly, number of primary care visits overall and yearly, number of mental and behavioral health encounters, number of dental visits overall and yearly, services received at visit
Change in type of preventive services received | 24 months prior to Medicaid expansion vs 24 months post
  Types of all billed encounters overall and yearly, number of primary care visits overall and yearly, number of mental and behavioral health encounters, number of dental visits overall and yearly, services received at visit
Change of Medicaid expenditures | 24 months prior to Medicaid expansion vs 24 months post
  The investigators will calculate the average pre-post expansion difference in total Medicaid expenditures. We will attach an expenditure for each service based on its average Medicaid Fee-For-Service reimbursement in the first year for those who were insured or uninsured pre or post expansion

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Marino M, Angier H, Fankhauser K, Valenzuela S, Hoopes M, Heintzman J, DeVoe J, Moreno L, Huguet N. Disparities in Biomarkers for Patients With Diabetes After the Affordable Care Act. Med Care. 2020 Jun;58 Suppl 6 Suppl 1(Suppl 6 1):S31-S39. doi: 10.1097/MLR.0000000000001257. PMID 32412951
- [Result] Marino M, Angier H, Springer R, Valenzuela S, Hoopes M, O'Malley J, Suchocki A, Heintzman J, DeVoe J, Huguet N. The Affordable Care Act: Effects of Insurance on Diabetes Biomarkers. Diabetes Care. 2020 Sep;43(9):2074-2081. doi: 10.2337/dc19-1571. Epub 2020 Jul 1. PMID 32611609
- [Result] Gemelas J, Marino M, Valenzuela S, Schmidt T, Suchocki A, Huguet N. Changes in diabetes prescription patterns following Affordable Care Act Medicaid expansion. BMJ Open Diabetes Res Care. 2021 Dec;9(Suppl 1):e002135. doi: 10.1136/bmjdrc-2021-002135. PMID 34933870
- [Result] Lindner SR, Marino M, O'Malley J, Angier H, Bailey SR, Hoopes M, Springer R, McConnell KJ, DeVoe J, Huguet N. Health Care Expenditures Among Adults With Diabetes After Oregon's Medicaid Expansion. Diabetes Care. 2020 Mar;43(3):572-579. doi: 10.2337/dc19-1343. Epub 2019 Dec 19. PMID 31857442
- [Result] Huguet N, Springer R, Marino M, Angier H, Hoopes M, Holderness H, DeVoe JE. The Impact of the Affordable Care Act (ACA) Medicaid Expansion on Visit Rates for Diabetes in Safety Net Health Centers. J Am Board Fam Med. 2018 Nov-Dec;31(6):905-916. doi: 10.3122/jabfm.2018.06.180075. PMID 30413546
- [Result] Angier H, Huguet N, Ezekiel-Herrera D, Marino M, Schmidt T, Green BB, DeVoe JE. New hypertension and diabetes diagnoses following the Affordable Care Act Medicaid expansion. Fam Med Community Health. 2020 Dec;8(4):e000607. doi: 10.1136/fmch-2020-000607. PMID 33334850
- [Result] Angier H, Ezekiel-Herrera D, Marino M, Hoopes M, Jacobs EA, DeVoe JE, Huguet N. Racial/Ethnic Disparities in Health Insurance and Differences in Visit Type for a Population of Patients with Diabetes after Medicaid Expansion. J Health Care Poor Underserved. 2019;30(1):116-130. doi: 10.1353/hpu.2019.0011. PMID 30827973
- [Derived] Hoopes M, Angier H, Raynor LA, Suchocki A, Muench J, Marino M, Rivera P, Huguet N. Development of an algorithm to link electronic health record prescriptions with pharmacy dispense claims. J Am Med Inform Assoc. 2018 Oct 1;25(10):1322-1330. doi: 10.1093/jamia/ocy095. PMID 30113681
- [Derived] Huguet N, Angier H, Marino M, McConnell KJ, Hoopes MJ, O'Malley JP, Raynor LA, Likumahuwa-Ackman S, Holderness H, DeVoe JE. Protocol for the analysis of a natural experiment on the impact of the Affordable Care Act on diabetes care in community health centers. Implement Sci. 2017 Feb 10;12(1):14. doi: 10.1186/s13012-017-0543-6. PMID 28183354